CLINICAL TRIAL: NCT01691833
Title: The Effect of Hypovitaminosis D and Vitamin D Supplementation on Fracture Nonunion Rates
Acronym: VitD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 01-11-09A
Record Dates: First submitted 2012-09-17; First posted 2012-09-25 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2018-10

CONDITIONS: Hypovitaminosis D
Keywords: Vitamin D; nonunion; long bone fracture; hypovitaminosis D
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vitamin D (Experimental): Patients that are deficient in Vitamin D will be assigned to the randomized arm of the study. They will be randomly chosen to receive either the Vitamin D supplement or the placebo.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Patients that are deficient in Vitamin D will be assigned to the randomized arm of the study. They will be randomly chosen to receive either the Vitamin D supplement or the placebo.
  Interventions: Dietary Supplement: Placebo
- Normovitaminosis (No Intervention): Patients with normovitaminosis( levels greater than or equal to 30ng/ml) will receive no intervention.

INTERVENTIONS:
Dietary Supplement: Vitamin D — Patients that are Vitamin D deficient and randomized to the treatment group will receive a 10,000 IU dose of Vitamin D.
  Arms: Vitamin D
Dietary Supplement: Placebo — Patients that are Vitamin D deficient maybe randomized to the placebo group D.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether vitamin D supplementation in patients with hypovitaminosis D can decrease nonunion (failure to heal) incidence in patients with fractures of the humerus, femur, or tibia. The central hypothesis of the study is that vitamin D supplementation in patients with fractures and hypovitaminosis D will decrease the risk of nonunion compared to placebo treatment.

DETAILED DESCRIPTION:
Vitamin D plays an important role in maintaining calcium and phosphate balance in the body and is important for maintenance of bone formation, remodeling, and healing. An extensive literature search indicates that although there is evidence that vitamin D deficiency is associated with fracture risk, there is no evidence of the role of vitamin D deficiency in subsequent failure to heal. The aims of study were to: 1) quantify the rate of hypovitaminosis D in an orthopedic trauma population in the Southeastern United States; 2) determine the rate of nonunion in vitamin D deficient patients, and 3) assess the feasibility of acute high-dose vitamin-D supplementation in hypovitaminosis D patients.

ELIGIBILITY:
Inclusion Criteria:

* presence of a long bone fracture (humerus, femur, or tibia)
* age greater than or equal to 18 years
* ability to follow-up at our clinic for 12 months

Exclusion Criteria:

* pathologic fractures (i.e. occuring in the presence of abnormal bone such as a tumor, cyst, or Paget's disease)
* open fractures (i.e. associated skin disruption) of Gustilo-Anderson type IIIB or C (i.e. significant soft-tissue and bone devitalization)
* presence of multiple fractures
* delay in presentation for initial treatment of more than 2 weeks from the time of injury
* preexisting disorders known to adversely affect bone healing (e.g. diabetes mellitus with HbA1C greater than or equal to 7, peripheral vascular disease, certain connective tissue disorders, and congenital or acquired disorders of bone metabolism)
* preexisting disorders affecting Vitamin D metabolism and/or calcium phosphate homeostasis (e.g. renal failure, hepatic failure, congenital defects in vitamin D metabolism, parathyroid disorders, conditions causing abnormal calcium and/or phosphate absorption)
* pregnant patients
* patients who are unable to provide consent for the study
* patients who are unable to swallow due to acuity of illness or physiologic reason
* prisoners who are patients because of their vulnerable population and inability to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-02; Primary Completion 2017-01 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Karunakar, MD, Principal Investigator — Wake Forest University Health Sciences; Rachel Seymour, PhD, Study Director — Wake Forest University Health Sciences; Christine Churchill, MA, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypovitaminosis- Vitamin D Group: Patients that are deficient in Vitamin D will be assigned to the randomized arm of the study. They will be randomly chosen to receive either the Vitamin D supplement or the placebo.
  Vitamin D: Patients that are Vitamin D deficient and randomized to the treatment group will receive a 10,000 IU dose of Vitamin D.
- Hypovitaminosis- Placebo Group: Patients that are deficient in Vitamin D will be assigned to the randomized arm of the study. They will be randomly chosen to receive either the Vitamin D supplement or the placebo.
  Placebo: Patients that are Vitamin D deficient maybe randomized to the placebo group D.
- Normovitaminosis: Patients with normovitaminosis D (levels greater than or equal to 30ng/ml) did not participate in the randomized portion of the study.
Period: Overall Study
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Started | 50 | 50 | 13
Completed | 49 | 49 | 13
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Normovitaminosis | Total
Number analyzed (Participants) | 50 | 50 | 13 | 113
Age, Customized [Mean (Standard Deviation); unit: years] | 38.9 (13.1) | 35.5 (12.1) | 39.9 (11.7) | 37.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 5 | 33
  Male | 34 | 38 | 8 | 80
Injury Type [Count of Participants; unit: Participants]
  Humerus | 8 | 7 | 3 | 18
  Femur | 25 | 25 | 5 | 55
  Tibia | 17 | 18 | 5 | 40
Tobacco use ( current) [Count of Participants; unit: Participants] | 24 | 23 | 8 | 55
BMI [Mean (Standard Deviation); unit: kg/m2] | 29.4 (6.3) | 27.8 (6.5) | 25.5 (4.87) | 28.3 (6.5)
Operatively treated [Count of Participants; unit: Participants] | 41 | 42 | 11 | 94
Prior use of Vitamins [Count of Participants; unit: Participants] | 29 | 36 | 6 | 71
Diabetes mellitus [Count of Participants; unit: Participants] | 0 | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Fracture Union
Description: Fracture Union is define as either clinical or radiological union. Clinical union defined as the absence of pain at the fracture site with the ability to bear full weight on the extremity without pain for activities of daily living (ambulation, lifting, carrying). Radiological union was determined by two blinded, independent review-ers and defined as the presence of bridging callus across at least three of four cortices or two of four cortices with a stable implant. When discrepancies between clinical and radiological union arose, the clinical assessment of union was preferred. Discrepancies in radiological outcomes were re-examined and a consensus view was obtained between reviewers if needed, to determine the outcome.If a patient did not meet the criteria for union and had at least nine months of follow•up or underwent re-operation for a diagnosis of a nonunion, they were deemed to have a nonunion.
Time Frame: up to 9 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Number analyzed (Participants) | 50 | 50 | 13
Participants | 40 | 39 | 10

2. Primary Outcome: Fracture Non-union
Description: If a patient did not meet the criteria for union and had at least nine months of follow-up or underwent re-operation for a diagnosis of a nonunion, they were deemed to have a nonunion.
Time Frame: 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Number analyzed (Participants) | 50 | 50 | 13
Participants | 2 | 2 | 3

3. Secondary Outcome: Fixation Failure
Description: Early failure of fixation was defined as the need to revise the fixation within three months.
Time Frame: three months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Number analyzed (Participants) | 50 | 50 | 13
Participants | 1 | 1 | 0

4. Secondary Outcome: Deep Infection
Description: A deep infection was defined as an unexpected return to theatre for irrigation and debridement with positive cultures from below the fascia.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Number analyzed (Participants) | 50 | 50 | 13
Participants | 0 | 1 | 0

5. Secondary Outcome: Lost to Follow-up
Description: Lost to follow-up if they did not meet the criteria for an outcome by 15 months after injury or surgery; were without another scheduled follow-up appointment, could not be contacted or refused to return for evaluation or send alternate records when contacted.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
Number analyzed (Participants) | 50 | 50 | 13
Participants | 7 | 7 | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Hypovitaminosis- Vitamin D Group | Hypovitaminosis- Placebo Group | Normovitaminosis
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/13
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No